CLINICAL TRIAL: NCT04913376
Title: Effectiveness of Hilotherapy for the Prevention of Oxaliplatin-induced Peripheral Neuropathy and Pain in the Treatment of Gastrointestinal Tumors: A Randomized Controlled Trial
Brief Title: Hilotherapy-study on Prevention of Oxaliplatin-induced Peripheral Neuropathy
Acronym: HILO-OXALI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S65284
Record Dates: First submitted 2021-05-06; First posted 2021-06-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Quality of Life; Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with stratification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hilotherapy (Experimental)
  Interventions: Device: Hilotherapy
- Standard care (No Intervention)

INTERVENTIONS:
Device: Hilotherapy — Constant cooling device for hands and feet.
  Arms: Hilotherapy

SUMMARY:
Effectiveness of hilotherapy for the prevention of oxaliplatin-induced peripheral neuropathy and pain in the treatment of gastrointestinal tumors: A randomized controlled trial.

DETAILED DESCRIPTION:
This study investigates whether constant cooling of the hands and feet using Hilotherm ChemoCare devices reduces the incidence of (severe) oxaliplatin-induced peripheral neuropathy and pain compared to standard care (i.e. no hand and foot cooling) in patients with gastrointestinal tumors.

ELIGIBILITY:
Most important Eligibility Criteria:

Inclusion Criteria:

* 18 years or older
* Gastro-intestinal tumor, treated in UZ Leuven (University Hospitals of Leuven)
* Starting oxaliplatin-based treatment

Exclusion Criteria:

* Already grade 2 or higher peripheral neuropathy

For a more detailed list, see protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Time until Grade 2 or higher patient-reported peripheral neuropathy after start of treatment in the first 12 weeks | 12 weeks
  Time-to-event analysis of Grade 2 or higher patient-reported peripheral neuropathy (severity scale, based on a patient-reported outcome questionnaire: "Patient-Reported Outcomes for Adverse Events" (PRO-CTCAE)). Outcome measurement value: percentage, absolute number, grade number.
  -- PRO-CTCAE: patient-reported outcome scale that assesses adverse events (e.g. "pain" and "numbness & tingling") on severity (5-point Likert scale 0 = "None", 1 = "Mild", 2 = "Moderate", 3 = "Severe", 4 = "Very severe") and interference with daily activities (0 = "Not at all", 1 = "A little bit", 2 = "Somewhat", 3 = "Quite a bit", 4 = "Very much"). We use the scale to assess the current experienced symptoms, and the scale has been translated to Dutch.

SECONDARY OUTCOMES:
Secondary Outcome Measures regarding peripheral neuropathy (pro-ctcae) | 24 weeks
  Time-to-event analysis and longitudinal analysis of a patient-reported outcome questionnaire (based on PRO-CTCAE: 4 items) and analysis of clinical decision-making to assess the incidence, severity and interference of peripheral neuropathy. Outcome measurement value: percentage, absolute number, grade number. This will be used to assess the cut-off point for the severity and interference experienced due to neuropathy.
Secondary Outcome Measures regarding peripheral neuropathy (eortc-qlq-cipn20) | 24 weeks
  Time-to-event analysis and longitudinal analysis of a PRO questionnaire (based on "European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Chemotherapy-induced Peripheral Neuropathy 20 items" (EORTC-QLQ-CIPN20)) and analysis of clinical decision-making to assess the incidence, severity and interference of peripheral neuropathy. Outcome measurement value: percentage, absolute number; to assess the degree of neuropathy in a more detailed way in comparison to the PRO-CTCAE.
  -- EORTC-QLQ-CIPN20: PRO scale that assesses 20 items (sensory (9), motor (8), autonomic symptoms (3)) with the use of a 4-point Likert scale (1 = "Not at all", 2 = "A little", 3 = "Quite a bit", 4 = "Very much"). We use the scale to assess the current experienced symptoms, and the scale has been translated to Dutch. Sum score will be calculated by item 1-18 (item 19: driving ability; item 20: male impotence; seperate assessment).
Secondary Outcome Measures regarding pain in hands and feet (pro-ctcae) | 24 weeks
  Time-to-event analysis and longitudinal analysis of a PRO questionnaire (based on PRO-CTCAE: 4 items) and analysis of clinical decision-making to assess the incidence, severity and interference of pain in hands and feet. Outcome measurement value: percentage, absolute number, grade number. This will be used to assess the cut-off point for the severity and interference experienced due to pain in hands and feet.
Secondary Outcome Measures regarding pain in hands and feet (eortc-qlq-cipn20) | 24 weeks
  Time-to-event analysis and longitudinal analysis of a PRO questionnaire (based on "European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire - Chemotherapy-induced Peripheral Neuropathy 20 items" (EORTC-QLQ-CIPN20)) and analysis of clinical decision-making to assess the incidence, severity and interference of pain in hands and feet. Outcome measurement value: percentage, absolute number; to assess the degree of pain in hands an feet in a more detailed way in comparison to the PRO-CTCAE.
Secondary Outcome Measures regarding comfort hilotherapy | 24 weeks
  Descriptive analysis of a patient-reported outcome questionnaire to assess comfort and compliance of hilotherapy. Outcome measurement value: percentage, absolute number. Self-developed 5-point Likert scale to assess patient experiences with three items: hilotherapy cuffs, tolerance of temperature and impact on mobility during chemotherapy (1 = "Very difficult", 2 = "Difficult", 3 = "Neutral", 4 = "Comfortable", 5 = "Very comfortable"), and one specific question regarding patient experiences with the impact of hilotherapy on their experiences of numbness & tingling and pain during the administration of hilotherapy (1 = "More severe", 2 = "Less severe", 3 = "Same experiences", 4 = "No present experiences of numbness & tingling and pain").

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Coolbrandt, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Flemish-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No